CLINICAL TRIAL: NCT05729607
Title: Vertical Soft Tissue Augmentation With Dermal Matrix and Enamel Matrix Derivative vs Connective Tissue Graft for the Treatment of Peri-implant Soft Tissue Dehiscences in the Esthetic Zone: A Randomized, Controlled, Clinical, Trial
Brief Title: Vertical Soft Tissue Augmentation With CTG vs ADM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Lorenzo Tavelli, Assistant Professor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITI IMP (22-0600)
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Implant Complication

STUDY DESIGN:
Intervention Model Description: Parallel-arm
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Connective tissue graft (Active Comparator): Autogenous connective tissue graft harvested from the palate as a free gingival graft and then de-epithelialized
  Interventions: Procedure: Vertical soft tissue augmentation
- Dermal matrix + EMD (Experimental): Acellular dermal matrix and enamel matrix derivative
  Interventions: Procedure: Vertical soft tissue augmentation

INTERVENTIONS:
Procedure: Vertical soft tissue augmentation — Vertical soft tissue augmentation with autogenous connective tissue graft (CTG)
  Arms: Connective tissue graft
Procedure: Vertical soft tissue augmentation — Vertical soft tissue augmentation with acellular dermal matrix (ADM) and enamel matrix derivative (EMD)
  Arms: Dermal matrix + EMD

SUMMARY:
The study aims at comparing two different approaches for vertical soft tissue augmentation at implant sites exhibiting soft tissue dehiscences: autogenous connective tissue graft vs acellular dermal matrix + enamel matrix derivative

DETAILED DESCRIPTION:
The present randomized clinical trial aims at investigating two approaches (autogenous connective tissue graft vs acellular dermal matrix + enamel matrix derivative) when performed for vertical soft tissue augmentation at sites with peri-implant soft tissue dehiscences. Clinical, volumetric, ultrasonographic, and patient-reported outcomes will be evaluated at different time points up to 1 year.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Periodontally and systemically healthy
* Full-mouth plaque score and full-mouth bleeding score ≤ 20% (measured at four sites per tooth)
* Presence of single functional dental implant in the anterior with a PSTD
* Implants diagnosed as healthy (Berglundh et al., 2018)

Exclusion criteria are:

* Contraindications for surgery
* Systemic condition (e.g. diabetes mellitus, HIV, cancer, etc) that could compromise wound healing
* Patients pregnant or attempting to get pregnant (self-reported)
* Untreated periodontitis
* Untreated peri-implant mucositis or peri-implantitis (Berglundh et al., 2018)
* Smoking, defined as self-reported daily habit. Occasional smokers won't be excluded
* History of soft tissue grafting at the implant site within the last 6 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2027-02-27 (Estimated); Study Completion 2027-11-27 (Estimated)

PRIMARY OUTCOMES:
Change in Soft tissue dehiscence depth | 12 months
  Change of the depth of the Soft tissue dehiscence (vertical measurement of the complication, in relation to the level of the cemento-enamel junction of the contralateral homologous tooth) at 12 months compared to baseline (expressed in millimeters)

SECONDARY OUTCOMES:
Complete peri-implant soft tissue dehiscence (PSTD) coverage | 12 months
  Percentage of cases with complete resolution of the implant esthetic complication (expressed as a percentage)
mean peri-implant soft tissue dehiscence (PSTD) coverage | 12 months
  Percentage of coverage of the soft tissue dehiscence compared to baseline, measured with a formula considering final PSTD depth and initial PSTD depth (expressed as a percentage)
Mucosal thickness changes | 3, 6, and 12 months
  Changes within the mucosal thickness measured with ultrasonography (expressed in mm)
3D Volumetric changes | 3, 6, and 12 months
  Changes within the buccal contour measured by superimposing digital impressions obtained with optical scanning (expressed in mm^3)
Post-operative pain | 14 days after the surgery
  Patient-reported pain after the surgical procedure (expressed with a 0-10 visual analogue scale [VAS])
Professional esthetic assessment (IDES) | 12 months
  Esthetic outcomes of the treatment assessed by a calibrated operator using the Implant soft tissue Dehiscence coverage Esthetic Score (IDES) (expressed using points, based on the IDES classification system from Zucchelli et al. 2021) The range is from 0 (worst outcome) to 10 (best outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Tavelli, DDS, MS, Principal Investigator — Harvard School of Dental Medicine, Boston, USA
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No